CLINICAL TRIAL: NCT00942162
Title: GSK2132231A Antigen-Specific Cancer Immunotherapeutic as First-line Treatment of Patients With Unresectable Metastatic Melanoma
Brief Title: A Study to Test the Benefit of a New Anti-cancer Treatment in Patients With Unresectable Advanced Melanoma
Acronym: PREDICT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111476; 2008-004007-64 (EudraCT Number)
Record Dates: First submitted 2009-07-09; First posted 2009-07-20 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Melanoma
Keywords: ASCI; Melanoma; Immunotherapeutic; Tumor antigen; PREDICT
MeSH Terms: conditions — Melanoma

ARMS (3):
- GSK2132231A GS+ Group (Experimental): Patients with the pre-specified gene signature (GS), who received intramuscularly up to 24 doses of MAGE-A3 ASCI (the study product), in 4 cycles. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening.
  Interventions: Biological: Immunotherapeutic GSK2132231A
- GSK2132231A GS- Group (Experimental): Patients without the pre-specified gene signature (GS), planned to receive intramuscularly up to 24 doses of MAGE-A3 ASCI (the study product), in 4 cycles. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening.
  Interventions: Biological: Immunotherapeutic GSK2132231A
- GSK2132231A GS-unknown Group (Experimental): Patients with unknown gene signature (GS), planned to receive intramuscularly up to 24 doses of MAGE_A3 ASCI (the study product), in 4 cycles. Gene-signature sub-grouping was based on patients having a potentially predictive gene signature, as assessed at screening.
  Interventions: Biological: Immunotherapeutic GSK2132231A

INTERVENTIONS:
Biological: Immunotherapeutic GSK2132231A — Intramuscular administration
  Other Names: MAGE-A3 ASCI

SUMMARY:
The objective of this study is to evaluate the clinical activity of the GSK2132231A immunotherapeutic in patients with MAGE-A3 positive unresectable metastatic melanoma presenting with the predictive gene signature.

DETAILED DESCRIPTION:
In this study, patients were to receive a maximum of 24 doses of recMAGE-A3 + AS15 according four cycles over a period of four years. An active follow-phase (up to five years after registration into the study) was planned for all patients.

As of Amendment 2, there will no longer be an active follow-up of patients after discontinuation or completion of the treatment. The study will end approximately 30 days after the last dose will be administered.

In addition, no more biological samples will be collected for protocol research purposes. For each biological sample already collected in the scope of this study and not tested yet, testing will not be performed by default, except if a scientific rationale remains relevant.

Blood sampling for safety monitoring as per protocol will continue.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with histologically proven metastatic cutaneous melanoma that is measurable.
* Patients with regional or distant cutaneous, subcutaneous or lymph-node metastasis can be included in the study, provided the disease is not amenable to curative treatment with surgery. In terms of the AJCC 2002 classification, this includes patients with unresectable stage III melanoma including in-transit metastases or patient with stage IV M1a melanoma.
* Written informed consent obtained from the patient prior to performance of any study specific procedure.
* Patient is >= 18 years at the time of signature of the informed consent form.
* The patient's tumor shows expression of MAGE-A3, as determined by RT-PCR analysis on a fresh tumor tissue sample obtained during the screening phase.
* Fresh tissue from the same lesion as used for MAGE-A3 expression testing must be available for the testing of the predictive gene signature.
* Formalin-fixed paraffin-embedded (FFPE) tissue must be available for complementary MAGE-A3 and gene signature testing.
* Patient fully recovered from any previous intervention (i.e., biopsy).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate bone-marrow reserve, adequate renal function and adequate hepatic function as assessed by standard laboratory criteria
* If the patient is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for at least 30 days prior to registration in the trial, have a negative pregnancy test and continue such precautions during the entire study treatment period and for 2 months after completion of the injection series.
* In the opinion of the investigator, the patient can and will comply with the protocol requirements.

Exclusion Criteria:

* Patients with unresectable stage IV M1b,c melanoma and patients with ocular and mucosal melanoma.
* The patient has at any time received any systemic anticancer treatment.
* Prior systemic treatment with an immunomodulator or loco-regional radiotherapy is permitted as prior adjuvant treatment provided that the last dose was administered at least 30 days before the registration into this trial;
* Previous adjuvant treatment with a cancer vaccine containing a tumor antigen other than MAGE-A3 is allowed if the last administration took place at least 8 weeks before registration into the trial.
* Prior isolated limb perfusion is permitted provided that the last dose was administered at least 30 days before registration into this trial
* The patient is scheduled to receive any anti-cancer specific treatment, including radiotherapy, other immunotherapy, chemotherapy and immunomodulating agents.
* The patient requires concomitant chronic treatment (more than 7 consecutive days) with systemic corticosteroids, or any other immunosuppressive agents.
* The patient has a history of autoimmune disease such as, but not limited to, multiple sclerosis, lupus, and inflammatory bowel disease. Patients with vitiligo are not excluded.
* The patient has a family history of congenital or hereditary immunodeficiency.
* The patient is known to be positive for Human Immunodeficiency Virus (HIV).
* History of allergic disease or reactions likely to be exacerbated by any component of the ASCI treatment.
* The patient has previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancer or carcinoma in situ of the cervix and effectively treated malignancy that has been in remission for over 5 years and is highly likely to have been cured.
* The patient has psychiatric or addictive disorders
* The patient has an uncontrolled bleeding disorder.
* The patient has concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
* Use of any investigational or non-registered product (drug or vaccine) other than the study medication within the 30 days preceding the first investigational treatment injection or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the patient has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device). For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2009-08-14 (Actual); Primary Completion 2012-06-27 (Actual); Study Completion 2015-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (60):
- United States (14):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Seattle, Washington
- France (11):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Boulogne
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Tours
- Germany (20):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Buxtehude, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Quedlinburg, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Erfurt, Thuringia
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
- Ireland (3):
  - GSK Investigational Site, Cork
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Galway
- Italy (4):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Siena, Tuscany
  - GSK Investigational Site, Padua, Veneto
- Poland (4):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=4962

REFERENCES:
- [Background] Saiag P, Gutzmer R, Ascierto PA, Maio M, Grob JJ, Murawa P, Dreno B, Ross M, Weber J, Hauschild A, Rutkowski P, Testori A, Levchenko E, Enk A, Misery L, Vanden Abeele C, Vojtek I, Peeters O, Brichard VG, Therasse P. Prospective assessment of a gene signature potentially predictive of clinical benefit in metastatic melanoma patients following MAGE-A3 immunotherapeutic (PREDICT). Ann Oncol. 2016 Oct;27(10):1947-53. doi: 10.1093/annonc/mdw291. Epub 2016 Aug 8. PMID 27502712
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 111476 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111476 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111476 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111476 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111476 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111476 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111476 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/ exclusion criteria, contraindications/ precautions, medical history of the patients and signing informed consent forms. While 125 subjects were enrolled, only 123 started the study, as 2 subjects did not receive treatment and were excluded.
Period: Overall Study
Arm/Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS-unknown Group
Started | 71 | 50 | 2
Completed | 1 | 0 | 0
Not Completed | 70 | 50 | 2
Not completed — Death | 45 | 35 | 0
Not completed — Withdrawal by Subject | 7 | 2 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Other | 14 | 13 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS-unknown Group | Total
Number analyzed (Participants) | 71 | 50 | 2 | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.9 (13.9) | 62.1 (12.6) | 60.5 (6.36) | 64.9 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 23 | 0 | 65
  Male | 29 | 27 | 2 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Caucasian/European heritage | 71 | 50 | 2 | 123

OUTCOME MEASURES:

1. Primary Outcome: One-year Overall Survival Rate (OSR) Estimated by Complete Case Method
Description: The 1-year overall survival rate (OSR) in the GS+ Population would be above 50% (target = 71%), a percentage which was reported together with its 95% confidence interval (CI). Maximum 1-year OSR of any currently available treatment in the MAGE-A3-positive population = 50% (P0). This median OS of 12 months is based on the observed median OS for MAGE-A3-positive patients, whose tumor did not present the predictive GS. The target 1-year OSR for patients presenting the predictive GS = 71% (P1). This corresponds to a median OS of 24 months when assuming an exponential distribution of OS.
Time Frame: Month 0 - Month 12
Population: The analysis was performed on the Total Treated Population (TTP), which included all patients who received at least one dose of study treatment, but did not include patients who dropped out from the study (i.e. patients alive at the last evaluation visit and followed for less than 1 year at first database freeze).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS-unknown Group
Number analyzed (Participants) | 65 | 48 | 2
Percentage of Participants | 83.08 [71.73 to 91.24] | 83.33 [69.78 to 92.52] | 100 [15.81 to 100.00]

2. Primary Outcome: Number of Patients Reported With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed included medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/ incapacity. Events which were part of the natural course of the disease under study (i.e., disease progression, recurrence) were captured as part of the clinical activity outcome variables in this study; therefore these did not need to be reported as SAEs. Progression/recurrence of the tumor in a patient was recorded as part of the clinical assessment data collection, and deaths due to progressive disease was recorded on a specific form, but not as an SAE. However, if the investigator considered that there was a causal relationship between treatment or protocol design/procedures and the disease progression/recurrence, then the event was reported as an SAE. Any new primary cancer (non-related to the cancer under study) was reported as an SAE.
Time Frame: Month 0 - Month 49
Population: The analysis was performed on the Total Treated Population (TTP), which included all patients who received at least one dose of study treatment. Safety was assessed in the overall population regardless of GS status.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Group: Group of all patients (GS+, GS- and Unknown GS) planned to receive intramuscularly up to 24 doses of MAGE-A3 ASCI (the study product), in 4 cycles.
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants | 19

3. Secondary Outcome: Number of Patients With Diseases Characteristics by GS
Description: Cancer staging (characteristics and categories) as by the categorization by the American Joint Committee on Cancer (AJCC) Staging Manual 2002: "Stage IIIA patients have up to three microscopic nodal metastases arising from a non-ulcerating primary melanoma and have an ' intermediate risk' for distant metastases and melanom-specific survival. Stage IIIB patients have up to three microscopic nodal metastases arising from a non-ulcerating melanoma or have up to three microscopic nodal metastases arising from an ulcerating melanoma, or have intralymphatic metastases without nodal metastases. They constitute a 'high-risk' group prognostically." The remaining patients with regional melanoma are Stage IIIC patients are at 'very high risk' for distant metastases and melanoma-specific mortality. Stage IV melanoma patients have metastasis at any distant site and constitute the group with the worst prognosis. Stage MC patients are those with confirmed missing cancer.
Time Frame: Month 0 - Month 49
Population: The analysis was performed on the Total Treated Population (TTP), which included all patients who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS-unknown Group
Number analyzed (Participants) | 71 | 50 | 2
Participants
  STAGE IIIA | 0 | 0 | 0
  STAGE IIIB | 11 | 4 | 1
  STAGE IIIC | 21 | 19 | 1
  STAGE IV | 39 | 27 | 0
  STAGE MC | 0 | 0 | 0

4. Secondary Outcome: Progression-free Survival (PFS) by GS
Description: From study start (Month 0) to Month 24, each patient was censored out of the analysis at 1st report of disease progression or death. PFS was defined and calculated as the time from first treatment to either the first progression of the disease or the date of death, whichever occurred first. In case a patient went off protocol treatment, the date of first documented progression (if applicable) was to be used as date of progression. Patients still alive with no evidence of disease progression at the time of their last visit or for whom date of first documented progression was not applicable, were censored at the time of the last examination. PFS analysis was performed using the non-parametric Kaplan-Meier method.
Time Frame: Month 0 - Month 24
Population: The analysis was performed on the Total Treated Population (TTP), which included all patients who received at least one dose of study treatment. PFS was not assessed in the MAGE-A3 Unknown GS Group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Overall Study Group | GSK2132231A GS+ Group | GSK2132231A GS- Group
Number analyzed (Participants) | 123 | 71 | 50
Months | 2.8 [2.8 to 2.8] | 2.8 [2.8 to 2.9] | 2.8 [2.5 to 2.8]

5. Secondary Outcome: Kaplan-Meier Estimates of the Progression-free Survival (PFS) at Months 6, 12 and 24, by Gene Signature
Description: PFS was defined as the time from the date of registration of the patient to either the date of disease progression or the date of death, whichever comes first. Patients alive and without disease progression were censored at the date of their last tumor evaluation. The PFS estimates were assessed by the Kaplan-Meier method and expressed as the percentage of patients who did not progress and were alive at a given time.
Time Frame: Month 6, Month 12, Month 24
Population: The analysis was performed on the Total Treated Population (TTP), which included all patients who received at least one dose of study treatment. PFS was not assessed in the GSK2132231A GS-unknown Group.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | GSK2132231A GS+ Group | GSK2132231A GS- Group
Number analyzed (Participants) | 71 | 50
Percentage of patients
  PFS 6M | 13.53 [6.71 to 22.75] | 5 [1 to 14.22]
  PFS 12M | 6.02 [1.95 to 13.43] | 5 [1 to 14.22]
  PFS 24M | 1.5 [0.13 to 7.12] | 5 [1 to 14.22]

6. Secondary Outcome: Overall Survival (OS) by GS
Description: OS was defined as the time from registration of the patient until death, with patients alive at the time of analysis censored at the time of the last contact.
Time Frame: Up to 5 years from the time of registration.
Population: The analysis was performed on the Total Treated Population (TTP), which included all patients who received at least one dose of study treatment. OS was not assessed in the GSK2132231A GS-unknown Group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Overall Study Group | GSK2132231A GS+ Group | GSK2132231A GS- Group
Number analyzed (Participants) | 123 | 71 | 50
Months | 23.9 [19.2 to 28.2] | 20.6 [16.1 to 28.2] | 25.8 [18.4 to 35.5]

7. Secondary Outcome: Time to Treatment Failure (TTF) by GS
Description: The TTF was defined as the time from registration of the patient until the date of the last treatment administration, irrespective of the reason for study treatment discontinuation.
Time Frame: Month 0 - Month 24
Population: The analysis was performed on the Total Treated Population (TTP), which included all patients who received at least one dose of study treatment. TTF was not assessed in the GSK2132231A GS-unknown Group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Overall Study Group | GSK2132231A GS+ Group | GSK2132231A GS- Group
Number analyzed (Participants) | 123 | 71 | 50
Months | 2.5 [2.4 to 4.1] | 2.7 [2.4 to 5.4] | 2.4 [2.3 to 2.6]

8. Secondary Outcome: Best Overall Response (BOR) by GS
Description: The BOR was the best response recorded from the start of the treatment until disease progression/ recurrence, except for confirmed objective response, which was reported as BOR independently of its time of occurrence. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI and/or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions without any new lesions and/or progression of existing non-target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (PD) without any new lesions and/or progression of existing non-target lesions; PD, >=20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; NE = Non-evaluable response.
Time Frame: Month 0 - Month 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS-unknown Group
Number analyzed (Participants) | 71 | 50 | 2
Participants
  CR | 0 | 1 | 0
  PR | 3 | 0 | 0
  SD | 11 | 4 | 0
  SD/ PR | 3 | 0 | 0
  PD | 51 | 44 | 2
  NE | 3 | 1 | 0
  Missing | 0 | 0 | 0

9. Secondary Outcome: Duration of Response (CR or PR)
Description: Duration of response was measured from the time when the measurement criteria for CR/ PR (whichever was recorded first) were met until the first date that recurrent or PD was objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started). Note: As there was only one patient analysed in the GSK2132231A GS- Group, the median duration of response was not calculated for this latter group.
Time Frame: Month 0 - Month 24
Population: The analysis was performed on the Responders Population, including patients with an objective response [complete (CR) or partial response (PR)] as best overall clinical response as confirmed by repeated assessments performed at least 4 weeks apart at the time of analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Overall Study Group | GSK2132231A GS+ Group | GSK2132231A GS- Group
Number analyzed (Participants) | 4 | 3 | 1
Months | 8.3 [1.9 to 8.3] | 6.9 [1.9 to 9.7] | NA [NA to NA] — Median duration of response cannot be calculated as number analyzed =1.

10. Secondary Outcome: Duration of Stable Disease (SD), or Time-to-Progression (TTP) by GS
Description: The duration of stable disease (SD), or TTP, was tabulated for patients whose best response was SD. The minimal time interval required between 2 measurements for determination of SD was 12 weeks.
Time Frame: Month 0 - Month 24
Population: The analysis was performed on the Stable Disease Population, which included the patients whose best response was stable disease. To qualify as SD for the best overall response, the patient should be in a SD status for a minimum of 12 weeks, as documented by two consecutive visits 12 weeks apart, or a SD status 12 weeks after baseline evaluation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Overall Study Group | GSK2132231A GS+ Group | GSK2132231A GS- Group
Number analyzed (Participants) | 15 | 11 | 4
Months | 5.4 [5.1 to 9.4] | 5.4 [4.1 to 9.4] | 5.4 [5.1 to 25]

11. Secondary Outcome: Number of Seropositive Patients for Anti-MAGE-A3
Description: Seropositive patients were those patients with anti-MAGE-A3 antibody concentrations ≥ 27 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: PRE = Pre any dose, PII(W4) = Post-Dose 2 (Week 4), PVI(W12) = Post-Dose 6 (Week 12), PXII(W31) = Post-Dose 12 (Week 31), PXVI(W54) = Post-Dose 16 (Week 54), PXVII(M18) = Post-Dose 17 (Month 18), PXXIV(M49) = Post-Dose 24 (Month 49).
Population: The analysis was performed on the According-To-Protocol Population (ATP) for immunogenicity, which included all evaluable patients for whom immunogenicity data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS-unknown Group
Number analyzed (Participants) | 87 | 52 | 34 | 1
Participants
  Anti-MAGE-A3, PRE | 7 | 4 | 3 | 0
  Anti-MAGE-A3, PII(W4): number analyzed (Participants) | 62 | 39 | 22 | 1
  Anti-MAGE-A3, PII(W4) | 60 | 37 | 22 | 1
  Anti-MAGE-A3, PVI(W12): number analyzed (Participants) | 52 | 34 | 17 | 1
  Anti-MAGE-A3, PVI(W12) | 52 | 34 | 17 | 1
  Anti-MAGE-A3, PXII(W31): number analyzed (Participants) | 11 | 5 | 6 | 0
  Anti-MAGE-A3, PXII(W31) | 11 | 5 | 6 | 0
  Anti-MAGE-A3, PXVI(W54): number analyzed (Participants) | 6 | 3 | 3 | 0
  Anti-MAGE-A3, PXVI(W54) | 6 | 3 | 3 | 0
  Anti-MAGE-A3, PXVII(M18): number analyzed (Participants) | 3 | 2 | 1 | 0
  Anti-MAGE-A3, PXVII(M18) | 3 | 2 | 1 | 0
  Anti-MAGE-A3, PXXIV(M49): number analyzed (Participants) | 4 | 4 | 0 | 0
  Anti-MAGE-A3, PXXIV(M49) | 4 | 4 | 0 | 0

12. Secondary Outcome: Anti-MAGE-A3 Antibody Concentrations
Description: Anti-MAGE-A3 antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in EL.U/mL.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Overall Study Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS-unknown Group
Number analyzed (Participants) | 87 | 52 | 34 | 1
EL.U/mL
  Anti-MAGE-A3, PRE | 11.2 [10.3 to 12.2] | 11.2 [10 to 12.5] | 11.3 [9.8 to 13] | 10.0 [NA to NA] — The limits of the CI can not be calculated as number analyzed =1.
  Anti-MAGE-A3, PII(W4): number analyzed (Participants) | 62 | 39 | 22 | 1
  Anti-MAGE-A3, PII(W4) | 906.1 [608 to 1350.2] | 728.7 [406 to 1307.9] | 1385.7 [896.4 to 2142] | 387.0 [NA to NA] — The limits of the CI can not be calculated as number analyzed =1.
  Anti-MAGE-A3, PVI(W12): number analyzed (Participants) | 52 | 34 | 17 | 1
  Anti-MAGE-A3, PVI(W12) | 6190.1 [5007.6 to 7652] | 5631 [4284.9 to 7399.8] | 7500.1 [5165.9 to 10889.2] | 5921.0 [NA to NA] — The limits of the CI can not be calculated as number analyzed =1.
  Anti-MAGE-A3, PXII(W31): number analyzed (Participants) | 11 | 5 | 6 | 0
  Anti-MAGE-A3, PXII(W31) | 6724.2 [3978 to 11366.4] | 7094.2 [2360 to 21325.5] | 6430.7 [2877.3 to 14372.4] |
  Anti-MAGE-A3, PXVI(W54): number analyzed (Participants) | 6 | 3 | 3 | 0
  Anti-MAGE-A3, PXVI(W54) | 3289.8 [1575.4 to 6870] | 2570.9 [480.1 to 13765.9] | 4209.7 [622.4 to 28473.7] |
  Anti-MAGE-A3, PXVII(M18): number analyzed (Participants) | 3 | 2 | 1 | 0
  Anti-MAGE-A3, PXVII(M18) | 4118.6 [1557.3 to 10892.7] | 4784.5 [115.5 to 198255.8] | 3052.0 [NA to NA] — The limits of the CI can not be calculated as number analyzed =1. |
  Anti-MAGE-A3, PXXIV(M49): number analyzed (Participants) | 4 | 4 | 0 | 0
  Anti-MAGE-A3, PXXIV(M49) | 7063.9 [3780.4 to 13199.4] | 7063.9 [3780.4 to 13199.4] |  |

13. Secondary Outcome: Number of Seropositive Patients for Protein D
Description: Seropositive patients were those patients with anti-PD antibody concentrations ≥ 100 EL.U/mL.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS-unknown Group
Number analyzed (Participants) | 88 | 53 | 34 | 1
Participants
  Anti-PD, PRE | 29 | 20 | 8 | 1
  Anti-PD, PII (W4): number analyzed (Participants) | 77 | 46 | 30 | 1
  Anti-PD, PII (W4) | 77 | 46 | 30 | 1
  Anti-PD, PVI (W12): number analyzed (Participants) | 52 | 34 | 17 | 1
  Anti-PD, PVI (W12) | 52 | 34 | 17 | 1
  Anti-PD, PXII (W31): number analyzed (Participants) | 11 | 5 | 6 | 0
  Anti-PD, PXII (W31) | 11 | 5 | 6 | 0
  Anti-PD, PXVI (W54): number analyzed (Participants) | 6 | 3 | 3 | 0
  Anti-PD, PXVI (W54) | 6 | 3 | 3 | 0
  Anti-PD, PXVII (M18): number analyzed (Participants) | 3 | 2 | 1 | 0
  Anti-PD, PXVII (M18) | 3 | 2 | 1 | 0
  Anti-PD, PXXIV (M49): number analyzed (Participants) | 4 | 4 | 0 | 0
  Anti-PD, PXXIV (M49) | 4 | 4 | 0 | 0

14. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD)
Description: Anti-PD antibody concentrations were presented as geometric mean concentrations (GMCs) and expressed in EL.U/mL.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Overall Study Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS-unknown Group
Number analyzed (Participants) | 88 | 53 | 34 | 1
EL.U/mL
  Anti-PD, PRE | 81.2 [68.5 to 96.2] | 86.1 [68.9 to 107.5] | 70.6 [54.5 to 91.5] | 412.0 [NA to NA] — The limits of the CI can not be calculated as number analyzed =1.
  Anti-PD, PII (W4): number analyzed (Participants) | 77 | 46 | 30 | 1
  Anti-PD, PII (W4) | 4588 [3397.5 to 6195.7] | 4196.9 [2768 to 6363.3] | 5139.8 [3253.3 to 8120.2] | 9167.0 [NA to NA] — The limits of the CI can not be calculated as number analyzed =1.
  Anti-PD, PVI (W12): number analyzed (Participants) | 52 | 34 | 17 | 1
  Anti-PD, PVI (W12) | 15036.7 [12057.7 to 18751.5] | 14091.9 [10763.7 to 18449.4] | 16453.2 [10607.9 to 25519.6] | 29553.0 [NA to NA] — The limits of the CI can not be calculated as number analyzed =1.
  Anti-PD, PXII (W31): number analyzed (Participants) | 11 | 5 | 6 | 0
  Anti-PD, PXII (W31) | 23548.6 [15167.2 to 36561.6] | 25070.5 [8468.5 to 74220] | 22351.2 [13378 to 37343.1] |
  Anti-PD, PXVI(W54): number analyzed (Participants) | 6 | 3 | 3 | 0
  Anti-PD, PXVI(W54) | 12389.9 [6229 to 24644.4] | 9639.2 [1286.9 to 72202.6] | 15925.5 [4872 to 52057] |
  Anti-PD, PXVII (M18): number analyzed (Participants) | 3 | 2 | 1 | 0
  Anti-PD, PXVII (M18) | 11386.1 [3141.7 to 41265.3] | 13839.4 [93.9 to 2040751] | 7707.0 [NA to NA] — The limits of the CI can not be calculated as number analyzed =1. |
  Anti-PD, PXXIV (M49): number analyzed (Participants) | 4 | 4 | 0 | 0
  Anti-PD, PXXIV (M49) | 10546.9 [1777.2 to 62591.1] | 10546.9 [1777.2 to 62591.1] |  |

15. Secondary Outcome: Anti-MAGE-A3 Antibody Response
Description: Anti-MAGE-A3 antibody response defined as: For initially seronegative patients: post-vaccination antibody concentration ≥ 27 EL.U/mL; For initially seropositive patients: post-vaccination antibody concentration ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: PII(W4) = Post-Dose 2 (Week 4), PVI(W12) = Post-Dose 6 (Week 12), PXII(W31) = Post-Dose 12 (Week 31), PXVI(W54) = Post-Dose 16 (Week 54), PXVII(M18) = Post-Dose 17 (Month 18), PXXIV(M49) = Post-Dose 24 (Month 49)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS-unknown Group
Number analyzed (Participants) | 62 | 39 | 22 | 1
Participants
  Anti-MAGE-A3, PII (W4) | 60 | 37 | 22 | 1
  Anti-MAGE-A3, PVI (W12): number analyzed (Participants) | 52 | 34 | 17 | 1
  Anti-MAGE-A3, PVI (W12) | 52 | 34 | 17 | 1
  Anti-MAGE-A3, PXII (W31): number analyzed (Participants) | 11 | 5 | 6 | 0
  Anti-MAGE-A3, PXII (W31) | 11 | 5 | 6 | 0
  Anti-MAGE-A3, PXVI (W54): number analyzed (Participants) | 6 | 3 | 3 | 0
  Anti-MAGE-A3, PXVI (W54) | 6 | 3 | 3 | 0
  Anti-MAGE-A3, PXVII (M18): number analyzed (Participants) | 3 | 2 | 1 | 0
  Anti-MAGE-A3, PXVII (M18) | 3 | 2 | 1 | 0
  Anti-MAGE-A3, PXXIV (M49): number analyzed (Participants) | 4 | 4 | 0 | 0
  Anti-MAGE-A3, PXXIV (M49) | 4 | 4 | 0 | 0

16. Secondary Outcome: Anti-PD Antibody Response
Description: Anti-PD antibody response defined as: For initially seronegative patients: post-vaccination antibody concentration ≥ 100 EL.U/mL; For initially seropositive patients: post-vaccination antibody concentration ≥ 2 fold the pre-vaccination antibody concentration.
Time Frame: as for outcome 15
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group | GSK2132231A GS+ Group | GSK2132231A GS- Group | GSK2132231A GS-unknown Group
Number analyzed (Participants) | 77 | 46 | 30 | 1
Participants
  Anti-PD, PII (W4) | 76 | 45 | 30 | 1
  Anti-PD, PVI (W12): number analyzed (Participants) | 52 | 34 | 17 | 1
  Anti-PD, PVI (W12) | 52 | 34 | 17 | 1
  Anti-PD, PXII (W31): number analyzed (Participants) | 11 | 5 | 6 | 0
  Anti-PD, PXII (W31) | 11 | 5 | 6 | 0
  Anti-PD, PXVI (W54): number analyzed (Participants) | 6 | 3 | 3 | 0
  Anti-PD, PXVI (W54) | 6 | 3 | 3 | 0
  Anti-PD, PXVII (M18): number analyzed (Participants) | 3 | 2 | 1 | 0
  Anti-PD, PXVII (M18) | 3 | 2 | 1 | 0
  Anti-PD, PXXIV (M49): number analyzed (Participants) | 4 | 4 | 0 | 0
  Anti-PD, PXXIV (M49) | 4 | 4 | 0 | 0

17. Secondary Outcome: Number of Patients With Abnormal Alanine Aminotransferase (ALT) Values by Maximum Grade
Description: The status of each patient as regards ALT laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G2, G3 and Unknown (UNK).
Time Frame: Month 0 - Month 49 (each patient was censored out of the analysis at time of death)
Population: The analysis was performed on the Total Treated Population (TTP), which included all patients who received at least one dose of study treatment and was assessed in the overall population regardless of GS status.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants
  ALT - SCR G0; SE G0 | 100
  ALT - SCR G0; SE G1 | 8
  ALT - SCR G0; SE G2 | 1
  ALT - SCR G0; SE G3 | 1
  ALT - SCR G0; SE UNK | 1
  ALT - SCR G1; SE G0 | 3
  ALT - SCR G1; SE G1 | 8
  ALT - SCR G1; SE G2 | 1

18. Secondary Outcome: Number of Patients With Abnormal Aspartate Aminotransferase (AST) Values by Maximum Grade
Description: The status of each patient as regards AST laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1 and Unknown (UNK).
Time Frame: Month 0 - Month 49 (each patient was censored out of the analysis at time of death)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants
  AST - SCR G0; SE G0 | 101
  AST - SCR G0; SE G1 | 12
  AST - SCR G0; SE UNK | 1
  AST - SCR G1; SE G0 | 6
  AST - SCR G1; SE G1 | 3

19. Secondary Outcome: Number of Patients With Abnormal Alkaline Phosphatase (ALK) Values by Maximum Grade
Description: The status of each patient as regards ALK laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1 and Unknown (UNK).
Time Frame: Month 0 - Month 49 (each patient was censored out of the analysis at time of death)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants
  ALK - SCR G0; SE G0 | 103
  ALK - SCR G0; SE G1 | 7
  ALK - SCR G0; SE UNK | 1
  ALK - SCR G1; SE G0 | 5
  ALK - SCR G1; SE G1 | 7

20. Secondary Outcome: Number of Patients With Abnormal Bilirubine (BIL) Values by Maximum Grade
Description: The status of each patient as regards BIL laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0), G1 and G2. CTC grade statuses reported at SE were G0, G1, G2 and Unknown (UNK).
Time Frame: Month 0 - Month 49 (each patient was censored out of the analysis at time of death)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants
  BIL - SCR G0; SE G0 | 113
  BIL - SCR G0; SE G1 | 5
  BIL - SCR G0; SE UNK | 1
  BIL - SCR G1; SE G0 | 2
  BIL - SCR G2; SE G1 | 1
  BIL - SCR G2; SE G2 | 1

21. Secondary Outcome: Number of Patients With Abnormal Creatinine (CREA) Values by Maximum Grade
Description: The status of each patient as regards CREA laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0), G1 and G2. CTC grade statuses reported at SE were G0, G1, G2 and Unknown (UNK).
Time Frame: Month 0 - Month 49 (each patient was censored out of the analysis at time of death)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants
  CREA - SCR G0; SE G0 | 105
  CREA - SCR G0; SE G1 | 7
  CREA - SCR G0; SE UNK | 1
  CREA - SCR G1; SE G0 | 1
  CREA - SCR G1; SE G1 | 6
  CREA - SCR G1; SE G2 | 2
  CREA - SCR G2; SE G2 | 1

22. Secondary Outcome: Number of Patients With Abnormal Hemoglobin (HGB) Values by Maximum Grade
Description: The status of each patient as regards HGB laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0), G1 and G2. CTC grade statuses reported at SE were G0, G1, G2, G3, G4, and Unknown (UNK).
Time Frame: Month 0 - Month 49 (each patient was censored out of the analysis at time of death)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants
  HGB - SCR G0; SE G0 | 61
  HGB - SCR G0; SE G1 | 30
  HGB - SCR G0; SE G2 | 1
  HGB - SCR G0; SE G3 | 1
  HGB - SCR G0; SE UNK | 1
  HGB - SCR G1; SE G0 | 1
  HGB - SCR G1; SE G1 | 16
  HGB - SCR G1; SE G2 | 6
  HGB - SCR G1; SE G3 | 3
  HGB - SCR G1; SE G4 | 1
  HGB - SCR G2; SE G0 | 1
  HGB - SCR G2; SE G2 | 1

23. Secondary Outcome: Number of Patients With Abnormal Leukocytes (LEU) Values by Maximum Grade
Description: The status of each patient as regards LEU laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0), G1 and G2. CTC grade statuses reported at SE were G0, G1, G2, G4, and Unknown (UNK).
Time Frame: Month 0 - Month 49 (each patient was censored out of the analysis at time of death)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants
  LEU - SCR G0; SE G0 | 99
  LEU - SCR G0; SE G1 | 10
  LEU - SCR G0; SE G2 | 1
  LEU - SCR G0; SE G4 | 1
  LEU - SCR G0; SE UNK | 1
  LEU - SCR G1; SE G0 | 6
  LEU - SCR G1; SE G1 | 3
  LEU - SCR G1; SE G2 | 1
  LEU - SCR G2; SE G1 | 1

24. Secondary Outcome: Number of Patients With Abnormal Lymphopenia (LYM) Values by Maximum Grade
Description: The status of each patient as regards LYM laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0), G1, G2 and G3. CTC grade statuses reported at SE were G0, G1, G2, G3 and Unknown (UNK).
Time Frame: Month 0 - Month 49 (each patient was censored out of the analysis at time of death)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants
  LYM - SCR G0; SE G0 | 67
  LYM - SCR G0; SE G1 | 18
  LYM - SCR G0; SE G2 | 3
  LYM - SCR G0; SE UNK | 1
  LYM - SCR G1; SE G0 | 3
  LYM - SCR G1; SE G1 | 23
  LYM - SCR G1; SE G2 | 4
  LYM - SCR G2; SE G2 | 1
  LYM - SCR G2; SE G3 | 1
  LYM - SCR G3; SE G3 | 2

25. Secondary Outcome: Number of Patients With Abnormal Neutrophils (NEU) Values by Maximum Grade
Description: The status of each patient as regards NEU laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0), G1 and G2. CTC grade statuses reported at SE were G0, G1, G2, G3 and Unknown (UNK).
Time Frame: Month 0 - Month 49 (each patient was censored out of the analysis at time of death)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants
  NEU - SCR G0; SE G0 | 108
  NEU - SCR G0; SE G1 | 4
  NEU - SCR G0; SE G2 | 1
  NEU - SCR G0; SE UNK | 1
  NEU - SCR G1; SE G0 | 2
  NEU - SCR G1; SE G1 | 5
  NEU - SCR G1; SE G3 | 1
  NEU - SCR G2; SE G1 | 1

26. Secondary Outcome: Number of Patients With Abnormal Platelets (PLT) Values by Maximum Grade
Description: The status of each patient as regards PLT laboratory values at baseline (SCR) up to study end (SE) was collected and graded according to the Common Terminology Criteria (CTC) Adverse event terminology, version 3.0. The post-treatment values were presented by worst grade versus baseline grade. SCR CTC grade statuses reported were Grade 0 (G0) and G1. CTC grade statuses reported at SE were G0, G1, G4, and Unknown (UNK).
Time Frame: Month 0 - Month 49 (each patient was censored out of the analysis at time of death)
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants
  PLT - SCR G0; SE G0 | 112
  PLT - SCR G0; SE G1 | 5
  PLT - SCR G0; SE G4 | 1
  PLT - SCR G0; SE UNK | 1
  PLT - SCR G1; SE G1 | 4

27. Secondary Outcome: Number of Patients With Autoimmune Diseases or Immune-mediated Inflammatory Disorders
Description: Auto-immune diseases or immune-mediated inflammatory disorders were tabulated during the whole duration of the study (up to 30 days after the last administration of the study treatment). The results were tabulated as Any event(s) reported.
Time Frame: Month 0 - Month 49
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants | 4

28. Secondary Outcome: Number of Patients Reported With Unsolicited Adverse Events (AEs) by Maximum Grade.
Description: The assessed AEs were ASCI-related adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE; Grade 5 = Death due to AE. An unsolicited AE covers any untoward medical occurrence in a clinical investigation patient temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Through 30 days after the last administration of the study treatment, approximately 49 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants
  Any event, Grade 1 | 52
  Any event, Grade 2 | 35
  Any event, Grade 3 | 21
  Any event, Grade 4 | 5
  Any event, Grade 5 | 3

29. Secondary Outcome: Number of Patients Reported With Unsolicited AE(s)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation patient temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Through 30 days after the last administration of the study treatment, approximately 49 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Group
Number analyzed (Participants) | 123
Participants | 116

ADVERSE EVENTS:
Time Frame: AEs were collected up to 30 days after each treatment; SAEs were collected from Month 0 to Month 49.
Description: As planned per study protocol, safety was assessed in the overall population regardless of GS status.
Arm/Group | Overall Study Group
All-Cause Mortality (participants affected / at risk) | 3/123
Serious Adverse Events (participants affected / at risk) | 19/123
Other Adverse Events (participants affected / at risk) | 107/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study Group (N=123)
Lymphoedema (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Atrial fibrillation (Cardiac disorders) | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Guillain-Barre syndrome (Nervous system disorders) | 1
Hypotonia (Nervous system disorders) | 1
Multi-organ failure (General disorders) | 1
Autoimmune colitis (Gastrointestinal disorders) | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Erysipelas (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study Group (N=123)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12)
Asthenia (General disorders) | 17 (42)
Chills (General disorders) | 21 (42)
Constipation (Gastrointestinal disorders) | 10 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Diarrhoea (Gastrointestinal disorders) | 13 (32)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (20)
Fatigue (General disorders) | 30 (110)
Headache (Nervous system disorders) | 14 (20)
Influenza like illness (General disorders) | 15 (46)
Injection site erythema (General disorders) | 21 (53)
Injection site pain (General disorders) | 60 (193)
Injection site reaction (General disorders) | 9 (38)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (96)
Nausea (Gastrointestinal disorders) | 15 (35)
Pain (General disorders) | 11 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (25)
Pyrexia (General disorders) | 41 (155)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.